CLINICAL TRIAL: NCT05513833
Title: Appalachian Specialty Telemedicine Access for Referrals (STAR) Trial
Brief Title: School Screening and Telemedicine Specialty Referral to Address Childhood Hearing Loss in Rural Kentucky
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: University of Kentucky (Other); Duke University (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 274089; 1U01OD033247 (NIH)
Record Dates: First submitted 2022-08-14; First posted 2022-08-24 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Hearing Loss
Keywords: Rural; hearing; loss; telemedicine; telehealth; school; disparities; screening
MeSH Terms: conditions — Hearing Loss | interventions — Referral and Consultation

STUDY DESIGN:
Intervention Model Description: 14 total counties (clusters) are participating in the stepped wedge randomized trial. There are two nested trials within the overall stepped-wedge trial: a complete design to evaluate the enhanced mHealth screening component and an incomplete design to evaluate the specialty telemedicine referral component combined with enhanced screening. Clusters will be randomized to cross over to enhanced mHealth hearing screening and specialty telemedicine referral in a stepwise manner until all clusters receive both the interventions.
  The enhanced mHealth screening component will be rolled out in Years 2 or 3 (control period in Years 1 and 2) depending on sequence randomization. Specialty telemedicine referral will be rolled out in Years 3 and 4 (control period in Years 2 and 3) depending on sequence randomization.
  Timeline update: With the trial extended by one year, rollout of specialty telemedicine referral will be shifted to Years 4 and 5 depending on sequence randomization.
Who Masked: Outcomes Assessor
Masking Description: Statisticians will also be masked to group allocation until analysis is complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): Standard School Screening: All counties in Sequence 1 will receive standard hearing screening in the control period, Year 1.
  Standard Referral: All counties in Sequence 1 will receive standard referral in control period, Years 1, 2, and 3, based on the updated timeline.
  Enhanced mHealth screening component: Counties randomized to Sequence 1 will receive the enhanced mHealth screening in Years 2, 3, 4, and 5, based on the updated timeline.
  Specialty telemedicine referral component: Counties randomized to Sequence 1 will receive the specialty telemedicine referral component in addition to the enhanced mHealth screening in Years 4 and 5, based on the updated timeline.
  Interventions: Other: Standard School Screening and Referral; Other: Enhanced mHealth Screening; Other: Specialty Telemedicine Referral
- Sequence 2 (Other): Standard Hearing Screening: All counties in Sequence 2 will receive standard hearing screening in the control period, Years 1 and 2.
  Standard Referral: All counties in Sequence 2 will receive standard referral in control period, Years 1, 2, 3, and 4, based on the updated timeline.
  Enhanced mHealth screening component: Counties randomized to Sequence 2 will receive the enhanced mHealth screening in Years 3, 4, and 5, based on the updated timeline.
  Specialty telemedicine referral component: Counties randomized to Sequence 2 will receive the specialty telemedicine referral component in addition to the enhanced mHealth screening in Year 5, based on the updated timeline.
  Interventions: Other: Standard School Screening and Referral; Other: Enhanced mHealth Screening; Other: Specialty Telemedicine Referral

INTERVENTIONS:
Other: Standard School Screening and Referral — Counties in the control condition will use standard hearing screening and standard referral by school district. Standard referral is typically a letter home from the school to parents/caregivers of children who refer screening.
Other: Enhanced mHealth Screening — The enhanced screening protocol will consist of an mHealth-based hearing screen combined with tympanometry.
Other: Specialty Telemedicine Referral — The specialty telemedicine referral will include a lay-friendly smartphone or tablet that connects to tools necessary for an ear and hearing evaluation. If a child requires referral from hearing screening, a school nurse/teacher will complete the established protocol for the specialty telemedicine referral and send details asynchronously to an audiologist for consultation.

SUMMARY:
This trial will evaluate a multilevel intervention (STAR model) that combines mobile health (mHealth) hearing screening tools with telemedicine technology for specialty care access in rural Kentucky schools. An initial version of the model was used in rural Alaska where telemedicine-based specialty referral improved both proportion of children receiving follow-up and time to follow-up. The refined STAR model will utilize an enhanced mHealth screening protocol that includes tympanometry for the detection of middle ear disease. The STAR model will also include a specialty telemedicine referral process in schools for children who refer school screening.

DETAILED DESCRIPTION:
Childhood hearing loss has substantial lifelong consequences, including speech-language delay, worse academic performance, and limited vocational opportunities. In rural settings, where access to care is limited, school-based preventative screening programs can help in early identification of childhood hearing loss. The state of Kentucky mandates hearing screening for all schools; however, the effectiveness of these programs is unclear. Further, current school programs do not include a middle ear assessment, which is needed to detect infection-related hearing loss common in children in rural and low-income settings. In children referred from school-based hearing screening programs, loss to follow-up also remains a pervasive issue.

To address these key issues, the University of Kentucky has partnered with the University of Arkansas Medical Sciences to lead the Appalachian STAR trial. This trial will evaluate a multilevel intervention (STAR model) that combines mobile health (mHealth) hearing screening tools with telemedicine technology for specialty care access in rural Kentucky schools. An initial version of the model was used in rural Alaska where telemedicine-based specialty referral improved both proportion of children receiving follow-up and time to follow-up. The refined STAR model will utilize an enhanced mHealth screening protocol that includes tympanometry for the detection of middle ear disease. The STAR model will also include a specialty telemedicine referral process in schools for children who refer school screening.

The Appalachian STAR stepped-wedge cluster randomized trial will be conducted in approximately 64 elementary schools located in 14 counties in rural Kentucky. Approximately 3600 students at school entry will be enrolled annually for 4 years, for a total of approximately 14,400 children. Cluster randomization will occur in two sequences at the county level, with 7 counties (clusters) in each sequence. The 4-year trial will include a control condition period, followed by phased roll-out of the intervention. The enhanced mHealth school hearing screening protocol will be implemented first. The following year, specialty telemedicine referral will be added to the enhanced screening protocol. All 14 counties will receive the STAR model by the end of the trial. An implementation evaluation will be conducted to refine the STAR model throughout the trial. If successful, the STAR model could be applied to address hearing loss and other childhood health conditions that affect underserved rural communities across America.

Timeline update: Based on feedback from community partners, we extended the trial for one year to allow for community-informed adaptations of the enhanced screening. After this additional year of enhanced screening only, specialty telemedicine referral will be added to the enhanced screening protocol. All counties will receive the STAR model by the end of the 5-year trial.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in school in one of the 14 participating counties
* Initial entry into elementary school
* Eligible regardless of age, gender, race, or ethnicity

Exclusion Criteria:

• N/A

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18000 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of children screened | School screening occurs once per school year, with timing and practices varying by school.
  This outcome will be measured at the end of each annual screening period for each school, for 5 years, based on the updated timeline.
Proportion of children who receive follow-up | Proportion of children who receive follow-up will be measured by the occurrence of an ear/hearing encounter, up to 60 days from the date of screening.
  This outcome will be measured each school year, for 3 years or 4 years depending on sequence randomization, based on the updated timeline.

CONTACTS AND LOCATIONS:
Overall Officials: Matt Bush, MD, PhD, MBA, Principal Investigator — University of Kentucky; Susan Emmett, MD, MPH, Principal Investigator — University of Arkansas Medical Sciences
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: Yes
This study focuses on population outcomes. School and health data will remain with local education and healthcare entities, and the study team will receive deidentified information. Data sharing will be considered upon request pending appropriate local approval.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Derived] Srinivasan T, Kleindienst Robler S, Turner E, Platt A, Arthur D, Prvu Bettger J, Lane H, Schuh Gebert M, Deshpande S, Schoenberg N, Bush ML, Emmett SD. Improving Access to Specialty Care for Rural Children Using Enhanced Hearing Screening and Specialty Telehealth Follow-Up in Rural Kentucky Schools: Protocol for a Hybrid Effectiveness-Implementation Stepped Wedge, Cluster-Randomized Controlled Trial (Appalachian STAR Trial). JMIR Res Protoc. 2025 Aug 26;14:e77630. doi: 10.2196/77630. PMID 40858294